CLINICAL TRIAL: NCT01046851
Title: Phase 3 Study of the Effects of Nopan as add-on Treatment to Antidepressants in Treating Depression and Suicidality
Brief Title: A Study of Nopan Treatment of Acute Suicidality
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Yoram Yovell (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Sponsor-Investigator, Prof. Yoram Yovell, MD, PhD, University of Haifa
Organization: University of Haifa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISAN-001-09
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2011-12

CONDITIONS: Suicidality
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nopan (Active Comparator)
  Interventions: Drug: Nopan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nopan — Nopan(0.2-1.6 mg/day, starting dose=0.2 mg/day, N=40)
  Other Names: Subotex
  Arms: Nopan
Drug: Placebo — Placebo in a manner similar to the active comparator
  Arms: Placebo

SUMMARY:
Anecdotal evidence and several clinical studies found the mixed opioid agonist-antagonist Nopan to be an effective antidepressant with a rapid onset of action. It is therefore hypothesized that Nopan may be a novel and quick-acting treatment for acute suicidality. Depression, suicidality, and overall functioning will be assessed before, during and after a four-week Nopan/placebo trial. It is hypothesized that subjects who receive the active drug will show rapid improvements in objective and subjective measures of these variables.

ELIGIBILITY:
Inclusion Criteria:

* suicidal behavior or ideation (BSI>6)

Exclusion Criteria:

* ECT history within the last month
* psychotic features within the last 3 months
* history of schizophrenia, substance or alcohol abuse within the last two years
* benzodiazepine dependence within the last two years
* any significant systemic illness or unstable medical condition which does not permit inclusion, according to the research physician
* pregnant women
* patients who currently suffer from severe impairment or severe dysfunction of liver, kidney, adrenal, gall, closed brain injury, urinary retention or respiratory system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in Suicidality as expressed by the score on the BSI | 4 weeks

SECONDARY OUTCOMES:
Reduction in depression as measured by the BDI | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Yovell, MD, PhD, Study Chair — University of Haifa, Institute for the Study of Affective Neuroscience; Mordechai Masiah, MD, Principal Investigator — Abarbanel MHC; Jack Asherov, MD, Principal Investigator — Edith Wolfson Medical Center; Nathaniel Laor, MD, PhD, Director, Principal Investigator — Tel Aviv- Brill Community Mental Health Center
Locations (3):
- Israel (3):
  - Abarbanel MHC, Bat Yam
  - Edith Wolfson Medical Center, Holon
  - Brill Community Mental Health Center, Tel Aviv